CLINICAL TRIAL: NCT05065710
Title: A Phase I, First-in-Human, Open-Label, Dose Escalation Study of ZL- 1211 in Patients With Unresectable or Metastatic Solid Tumor
Brief Title: A Study of ZL-1211 in Patients With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zai Biopharmaceutical (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZL-1211-001
Record Dates: First submitted 2021-09-12; First posted 2021-10-04 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumor
Keywords: CLDN18.2; Solid tumor

STUDY DESIGN:
Intervention Model Description: Phase I, the Dose Escalation Phase of the study will enroll patients with locally advanced or metastatic solid tumors of any histology with positive CLDN18.2. Phase II, the Cohort Expansion Phase of the study, will be conducted after determination of the dose level (RP2D) for cohort expansion based on the results of Phase I to explore the preliminary efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZL-1211 monotherapy (Experimental)
  Interventions: Drug: ZL-1211

INTERVENTIONS:
Drug: ZL-1211 — Phase 1 dose escalation part will enroll about 12-42 patients, Phase 2 dose expansion part will enroll about 15-40 patients in each cohort

SUMMARY:
This study is a Phase I/II, open-label, dose escalation, and cohort expansion study designed to characterize the safety, tolerability, pharmacokinetic (PK), pharmacodynamics (PD), immunogenicity, and preliminary antitumor activity of ZL-1211 administered by IV infusion on a every 2 weeks (Q2W) schedule.

DETAILED DESCRIPTION:
The study consists of two stages, Phase I -Dose Escalation Phase to determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) (if no MTD is defined) of ZL-1211, and Phase II -Cohort Expansion Phase to further define the safety and initial antitumor activity of ZL-1211 with the dose established in the Dose Escalation Phase. The trial was intended to be a Phase 1/2 trial but the Phase 2 was not initiated.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if all the following inclusion criteria apply:

1. Adults≥ 18 years of age.
2. Willing and able to provide signed and dated informed consent prior to any study related procedures and willing and able to comply with all study procedures.
3. All patients from Phase I and Phase II are required to provide tumor tissue for CLDN18.2 IHC assessment, and only patients with CLDN18.2-positive tumors will be included in this study.
4. Patients with histologically or cytologically confirmed metastatic or locally advanced solid tumors, refractory to standard treatment
5. Evaluable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Adequate hepatic function

   1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN).
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; AST or ALT ≤ 5 × ULN if liver metastases are present.
8. Adequate renal function, as defined by serum creatinine < 1.5 × ULN OR calculated creatinine CL > 40 mL/min, Cockroft-Gault Equation:
9. Hematological function defined as:

   1. Absolute neutrophil count ≥ 1.5 × 109/L without growth factor support in the 2 weeks prior to screening.
   2. Platelet count ≥ 100 × 109/L without transfusion in the 2 weeks prior to screening.
   3. Hemoglobin ≥ 9 g/dL without transfusion in the 2 weeks prior to screening.
10. Prothrombin time, international normalized ratio or/and activated partial thromboplastin time < 1.5 × ULN.
11. Recovery, to Grade 0-1, from AEs related to prior anticancer therapy except alopecia, < Grade 2 sensory neuropathy, lymphopenia.

Exclusion Criteria:

1. Patient with known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome related illness or known active or chronic hepatitis B virus infection or hepatitis C virus.
2. Any uncontrolled active infection.
3. Previous exposure to any CLDN18.2 antibody or CLDN18.2 chimeric antigen receptor T cell therapy.
4. Newly diagnosed or symptomatic brain metastases anticonvulsants are allowed.
5. Severe cardiovascular disease; New York Heart Association Class II-IV heart failure within 6 months of screening; uncontrolled arrhythmia within 6 months of screening.
6. Anticancer therapy or radiation therapy within 5 half-lives or 4 weeks (whichever is shorter) prior to screening; palliative radiotherapy within 2 weeks prior to screening.
7. Major surgery within 4 weeks prior to first dose; minor surgery within 2 weeks prior to first dose.
8. Symptomatic intrinsic lung disease (chronic obstructive pulmonary disease, pulmonary fibrosis).
9. Gastrointestinal abnormalities including:

   1. Documented unresolved gastric outlet obstruction or persistent vomiting defined as ≥ 3 episodes within 24 hours.
   2. Active peptic ulcer disease required treatment in the past 3 months.
   3. Gastrointestinal bleeding as evidenced by hematemesis, hematochezia, or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy.
   4. Documented active colitis within 4 weeks prior to study entry, including infectious colitis, radiation colitis and ischemic colitis.
   5. History of ulcerative colitis or Crohn's disease.
10. Patient has received systemic immunosuppressive therapy, including systemic corticosteroids 2 weeks prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-03-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Phase I ：MTD or MAD | One month
  To determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) (if no MTD is defined) of ZL-1211
Phase I and Phase II: safety and tolerability | Approximately 10 months
  Incidence of Treatment-Related Adverse Events as Assessed by CTCAE v5.0
Phase II: preliminary antitumor activity | Approximately 10 months
  Objective response rate defined as the proportion of patients with partial response (PR) proportion of patients with partial response (PR) or complete response (CR) based on Investigator assessment of tumor lesions per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Phase I and Phase II: pharmacokinetics (PK):AUC | Approximately 10 months
  Area under the curve (AUC)
Phase I and Phase II: pharmacokinetics (PK):Cmax | Approximately 10 months
  Maximum serum concentration (Cmax)
Phase I and Phase II: pharmacokinetics (PK):Tmax | Approximately 10 months
  Time to reach Cmax (Tmax)
Phase I and Phase II: pharmacokinetics (PK):Ctrough | Approximately 10 months
  Ctrough
Phase I and Phase II: pharmacokinetics (PK):Vss | Approximately 10 months
  Volume of distribution at steady state (Vss)
Phase I and Phase II: pharmacokinetics (PK):CL | Approximately 10 months
  Clearance (CL)
Phase I and Phase II: pharmacokinetics (PK):t1/2 | Approximately 10 months
  Half-life (t1/2)
Phase I and Phase II: immunogenicity | Approximately 10 months
  Incidence of anti-drug antibodies (ADAs)
Phase I and Phase II: immunogenicity | Approximately 10 months
  Quantity of anti-drug antibodies (ADAs)
Phase II: preliminary antitumor activity | Approximately 10 months
  Duration of response (DOR), defined as the time from the first date of objective response (CR or PR) to the first documented date of disease progression per RECIST v1.1 or the date of death due to any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (21):
- United States (10):
  - Zai Lab Site 2012, Scottsdale, Arizona
  - Zai Lab Site 2016, Lynwood, California
  - Zai Lab Site 2014, Indianapolis, Indiana
  - Zai Site 2020, Hackensack, New Jersey
  - Zai Lab Site 2025, New York, New York
  - Zai Lab Site 2015, Cincinnati, Ohio
  - Zai Lab Site 2011, Nashville, Tennessee
  - Zai Lab Site 2023, Fairfax, Virginia
  - Zai Lab Site 2013, Spokane, Washington
  - Zai Lab Site 2022, Tacoma, Washington
- China (11):
  - Zai Lab Site 1725, Hefei, Anhui
  - Zai Lab Site 1548, Beijing, Beijing Municipality
  - Zai Lab Site 1551, Harbin, Heilongjiang
  - Zai Lab Site 1549, Zhengzhou, Henan
  - Zai Lab Site 1202, Zhengzhou, Henan
  - Zai Lab Site 1537, Wuhan, Hubei
  - Zai Lab Site 1539, Jinan, Shandong
  - Zai Lab Site 1542, Shanghai, Shanghai Municipality
  - Zai Lab Site 1712, Chengdu, Sichuan
  - Zai Lab Site 1529, Hangzhou, Zhejiang
  - Zai Lab Site 1714, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Konno H, Lin T, Wu R, Dai X, Li S, Wang G, Chen M, Li W, Wang L, Sun BC, Luo Z, Huang T, Chen Y, Zhang J, Ye Q, Bellovin D, Wan B, Kang L, Szeto C, Hsu K, Kabbarah O. ZL-1211 Exhibits Robust Antitumor Activity by Enhancing ADCC and Activating NK Cell-mediated Inflammation in CLDN18.2-High and -Low Expressing Gastric Cancer Models. Cancer Res Commun. 2022 Sep 7;2(9):937-950. doi: 10.1158/2767-9764.CRC-22-0216. eCollection 2022 Sep. PMID 36922936